CLINICAL TRIAL: NCT03855657
Title: Investigating the Intestinal Microbiota, Epigenetic Markers and Body Fluid Metabolites to Identify Biomarkers for Inflammatory Bowel Diseases
Brief Title: Biobank - Investigating the Gut Microbiota, Genetics, Epigenetics and Metabolites
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: IBD Biobank Study
Record Dates: First submitted 2018-06-27; First posted 2019-02-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Biobank
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Stool, Saliva and biopsies from gastrointestinal tract
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inflammatory Bowel Disease Patient: Patient with confirmed diagnosis of Inflammatory Bowel Disease
- Healthy control: Controls (non-IBD) will comprise individuals undergoing colonoscopy for polyp or colorectal cancer screening, or investigations of gastrointestinal symptoms, and friends and spouses or partners of patients at Prince of Wales Hospital or Alice Ho Miu Ling Nethersole Hospital, or any individuals who are interested to participate in this study.
- Healthy relatives of Inflammatory Bowel Disease patient: Relatives or household members of both patients with IBD or other diseases and controls will be recruited.

SUMMARY:
Inflammatory bowel disease (IBD) affects 1 in 500 to 1,000 people in the West. Previously a disease predominantly of the West, there is now a marked increase in the incidence of ulcerative colitis (UC) and Crohn's disease (CD) in Asia, with an estimated prevalence of 1 in 3,000 and 1 in 10,000 respectively[1]. The rapid increase of IBD in Asian raising concern of investigators. Therefore setting up a large scale biobank with comprehensive clinical data is require.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) affects 1 in 500 to 1,000 people in the West. Previously a disease predominantly of the West, there is now a marked increase in the incidence of ulcerative colitis (UC) and Crohn's disease (CD) in Asia, with an estimated prevalence of 1 in 3,000 and 1 in 10,000 respectively [1]. IBD is thought to result from an aberrant immune response to intestinal bacteria in genetically susceptible individuals [2]. Genetic variants have been shown to contribute to an increased IBD risk. Although genetic traits predispose to the development of IBD in Asia, the change in epidemiology that has occurred over only a few decades suggests that other, presumably environmental factors play the major role in the development of disease [10].

IBD patients often rely on medical therapy to achieve remission. Due to the diverse features of severity, phenotypes, clinical courses and responses, personalizing IBD therapy is important to maximize management efficacy, minimize adverse events and decrease cost. Thiopurines is a key component of medications in the treatment of Inflammatory Bowel Disease (IBD). However, achieving an optimal efficacious thiopurine dosing can be difficult, as up to 10% of patients have dose-dependent toxicities and up to 9% of patients are resistant to thiopurine therapy [16, 17]. Such clinical toxicity could be due to inherited genetic variation of certain enzyme, leading to an unusual metabolic pathway, which generates toxic metabolites. On the other hand, few studies have studied the longitudinal changes in the gut microbiome with drug treatment in IBD. Shaw et al. characterized 19 children with CD and 4 with ulcerative colitis (UC), showing that dysbiosis at baseline correlated with the degree of inflammatory burden of luminal disease.Therefore, identification of comprehensive targets for drug monitoring will improve our understanding of the basis for inter-patient variability in drug toxicity and efficacy, and enable more individualized therapy.

Metabolism has an essential role in biological systems; and metabolites represent the end products of this important process from a cell of a certain physiological status. Blood and urine are integrative fluids that incorporates the metabolic outputs at different of the body, and thus providing a metabolic footprint as an end product [4].

Metagenomics which is a study of microbes as communities is also an important approach to study microbiota in human.The interplay between microbiota and genetics gives unique transcription profiles in the gut, and gene expression analyses provide insights into the transcriptional activity and functional molecular pathways underlying disease progression. Therefore, deep sequencing analysis of the colon suggests hypotheses about the pathophysiological processes in IBD patients. Further transcriptomics study and in combination with other meta'omics studies will provide the basis for in-depth understanding of IBD pathogenesis.

Due to the bio-clinical complexity of diseases and microbiota, a long term, large-scale prospective biobank is necessary to carry out meaningful research. This biobank will provide a powerful platform for studying a range of complex factors associated with IBD that are of great relevance to public health. Such biobank may be extended to other diseases including GI diseases and autoimmune disorder, which may possibly provide insight to the role of microbiota in human health.

In conclusion, a comprehensive understanding of the intestinal ecosystem, epigenetic, metabolic and transcription profiles, as well as their mechanisms in the disease pathogenesis in patients with IBD and other diseases may help us identify potential biomarkers. However, our current knowledge about them is still very limited, particularly in Asian patients, who have not been extensively researched. Further investigation in this field is needed. To serve these purposes, we aim to setup a large scale biobank with comprehensive clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 with a diagnosis of Crohn's disease or ulcerative colitis
* Informed Consent obtained

Exclusion Criteria:

* Known current infection with an enteric pathogen
* Previously been diagnosed with IBD (Control)
* Have a first of second degree relative with IBD (Control)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Crohn's disease or ulcerative colitis defined by endoscopy, radiology and histology
  Control will comprise individuals undergoing colonoscopy for polyp or colorectal cancer screening, or investigations of gastrointestinal symptoms, and friends and spouses or partners of patients at Prince of Wales Hospital or Alice Ho Miu Ling Nethersole Hospital, or any individuals who are interested to participate in this study.
  Relatives or household members of both patients with IBD or other diseases and controls will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2034-02 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
Setup a large scale biobank | 20 years
  Set up a large scale biobank to collect data such as comprehensive clinical data, such as patient's demographic and clinical information (e.g. age, weight, gender, family history of IBD, appendectomy history, drug usage etc.)

SECONDARY OUTCOMES:
Intestinal microbiota of IBD patient | 20 years
  Study samples will be collected to characterize which microbiota affect severity of IBD by performing metagenomics of gut microbiome in stool and biospy samples
Genetics and epigenetic markers in IBD | 20 years
  Study samples will be collected from patients with IBD and other diseases for genetic material isolation and gene expression checking by performing PCR.
Therapeutic drug monitoring | 20 years
  To understand the metabolic pathway leading to the target metabolites and therapeutic drug monitoring during following up by filling in questionniare
Biomarker of IBD | 20 years
  Study samples will be collected to characterize which microbiota affect severity of IBD by performing metagenomics of gut microbiome in stool and biospy samples
Pathobionts of IBD | 20 years
  Study samples will be collected to identify specific pathobionts that induce innate immune response by analysis of laboratory result (e.g. cell tissue culturing analysis of specific toxin to cells etc.)
Microbiota-induced molecular mechanisms | 20 years
  Study samples will be collected to characterize which Microbiota-induced molecular mechanisms by performing metagenomics of gut microbiome in stool and biospy samples
Disease pathogenesis | 20 years
  Study samples will be collected to characterize which microbiota induces disease by performing metagenomics of gut microbiome in stool and biospy samples

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong